CLINICAL TRIAL: NCT02905916
Title: The Efficacy and Safety of PEG-rhG-CSF in Neutropenia After Chemotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSPC-JYL-05-07
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Mammary Cancer; Lymphoma; Bone Tumour; Gynecological Tumors
MeSH Terms: conditions — Breast Neoplasms; Lymphoma; Bone Neoplasms | interventions — pegylated granulocyte colony-stimulating factor

ARMS (1):
- PEG-rhG-CSF (Experimental)
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF

SUMMARY:
The purpose of the trail is to evaluate the efficacy and safety of PEG-rhG-CSF in primary prophylaxis and secondary prophylaxis of neutropenia after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age between 18 and 70 years.
2. Breast cancer, lymphoma, bone tumor or Gynecologic tumor patients.
3. With multi-cycle chemotherapy.
4. With III/IV degree neutropenia after the last cycle of chemotherapy and plans to use the same regimen in the subsequent cycles.FN risk of the chemotherapy regimens is ≥20%，or 10%≤FN risk<20% and has high risk factors associated with FN.
5. KPS score≥ 70.
6. Expected to survive more than 3 months.
7. No hematologic system disease and ANC≥1.5×10E9/L, PKT≥80×10E9/L, Hb≥ 75g/L, WBC≥3×10E9/L, and no bleeding tendency.
8. Written informed consent are acquired. -

Exclusion Criteria:

1. With infection or systemic antibiotic therapy 72h before chemotherapy.
2. With any abnormal hematopoietic function.
3. Received transplantation within 3 months.
4. Suffered from other malignant tumor or brain metastases.
5. TBIL, ALT,AST > 2.5×ULN; if it were caused by liver metastases, TBIL, ALT,AST >5×ULN.
6. Cr >1.5 ×ULN.
7. Sensitive to the product or other genetically engineered biological products from Escherichia coli strains.
8. Mental or nervous system disorders.
9. Refused to accept contraceptive measures.
10. Other situations that investigators consider as contra-indication for this study.

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of febrile neutropenia (FN) | 30days after PEG-rhG-CSF administration

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, China